CLINICAL TRIAL: NCT05317845
Title: A Multi-center, Cross-sectional Chart Review and Survey to Capture the Prevalence and Clinical Management of Atherosclerotic Cardiovascular Diseases in Patients With Type 2 Diabetes Across Countries in the Middle East and Africa
Brief Title: An International Chart Review and Survey for the Prevalence and Clinical Management of Atherosclerotic Cardiovascular Diseases in Patients With Type 2 Diabetes Across Countries in the Middle East and Africa
Acronym: PACT-MEA
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-007; U1111-1266-5511 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Type 2 Diabetes (T2D): Selected for inclusion in the study by their primary or secondary care physicians
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — The clinical management and prescribed treatment of diabetes and eASCVD/ASCVD risk factors are independent of this study and are part of the routine clinical practice at the discretion of the treating physician.

SUMMARY:
The study is intended to estimate the proportion and clinical management of people with type 2 diabetes having atherosclerotic cardiovascular diseases or who are at high risk to develop atherosclerotic cardiovascular diseases.

Participants will be asked to give information about their health. Partipants will continue normal way of life and will not get any medication other than those prescribed to them by the doctor.

The study will last for about 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age greater than or equal to 18 years at the time of signing informed consent.
3. Diagnosed with T2D grater than or equal to 180 days prior to the day of signing informed consent

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Mental incapacity, unwillingness, inability, or language barriers precluding adequate understanding or cooperation
3. Diagnosed with Type 1 Diabetes (T1D).
4. Patients with known congenital heart disease/malformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetes (T2D) patients seen in routine visits
Sampling Method: Non-Probability Sample
Enrollment: 4089 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Established Atherosclerotic Cardiovascular Disease (eASCVD) pooled across all countries and separately for each country in scope | At the time of patient enrolment (Day 1)
  Percentage patients

SECONDARY OUTCOMES:
Proportion of T2D patients with high risk of Atherosclerotic cardiovascular disease (ASCVD) and without eASCVD | At the time of patient enrolment (Day 1)
  Percentage patients

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (7):
- Novo Nordisk Investigational Site, Manama, Bahrain
- Novo Nordisk Investigational Site, Alexandria, Egypt
- Novo Nordisk Investigational Site, Amman, Jordan
- Novo Nordisk Investigational Site, As Sālimīyah, Kuwait
- Novo Nordisk Investigational Site, Doha, Qatar
- Novo Nordisk Investigational Site, Johannesburg, South Africa
- Novo Nordisk Investigational Site, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Verma S, Sabbour H, Alamuddin N, Alawadi F, Alkandari H, Almahmeed W, Assaad-Khalil SH, Haddad J, Lombard L, Malik RA, Mashaki Ceyhan E, Prasad P, Tombak G, Salek S. A cross-sectional study of the prevalence and clinical management of atherosclerotic cardiovascular diseases in patients with type 2 diabetes across the Middle East and Africa (PACT-MEA): Study design and rationale. Diabetes Obes Metab. 2023 Jun;25(6):1444-1452. doi: 10.1111/dom.15011. Epub 2023 Mar 3. PMID 36775980
- [Derived] Salek S, Sabbour H, Alamuddin N, Alawadi F, Alkandari H, Almahmeed W, Assaad-Khalil SH, Ceyhan EM, Haddad J, Lombard L, Ngome M, Malik RA, Yadav G. Physician self-reported factors driving clinical decision-making in management of patients with T2D and ASCVD/high risk of ASCVD across the middle East and Africa: a cross-sectional study. Front Pharmacol. 2025 Sep 9;16:1558515. doi: 10.3389/fphar.2025.1558515. eCollection 2025. PMID 40994644
- [Derived] Assaad-Khalil SH, Bassyouni A, Toaima D, Gawish HS, El Hefnawy H, Megallaa M, Abushady M, ElKafrawy N, Hosny SS, Massoud TM. Prevalence and risk factors of atherosclerotic cardiovascular disease in Egyptians with type 2 diabetes: findings from the PACT-MEA study and call for action. BMJ Open. 2025 Aug 3;15(8):e092861. doi: 10.1136/bmjopen-2024-092861. PMID 40754331
- [Derived] Haddad JA, Annabi FOA, Abbasi H, AlSamen MAA, Ammari FL, Haddad FH, Haddad SE, Jaradat M, Khassawneh A, Khatib N, Magableh A, Al-Mousa E. The Prevalence of Atherosclerotic Cardiovascular Disease in Patients with Type 2 Diabetes in Jordan: The PACT-MEA Study. Diabetes Ther. 2025 May;16(5):899-913. doi: 10.1007/s13300-025-01718-7. Epub 2025 Mar 19. PMID 40106223